CLINICAL TRIAL: NCT04159233
Title: Pilot Study: Developing A Scalable Sleep Health Intervention to Improve Pain, Quality of Life, and Health in Former NFL Players
Brief Title: Sleep Bootcamp: A Pilot Tele-Sleep Program for Former National Football League (NFL) Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Principal Investigator, Suzanne M. Bertisch, MD, MPH, Assistant Professor, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019P002027
Record Dates: First submitted 2019-10-29; First posted 2019-11-12 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Sleep; Insomnia; Pain; Quality of Life
Keywords: sleep; pain; professional athlete; National Football League; Behavioral intervention
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adapted 'Brief Behavioral Therapy for Insomnia' (BBTI) (Other): All participants will receive the same intervention in this pilot study.
  Interventions: Behavioral: Brief Behavioral Therapy for Insomnia (BBTI)

INTERVENTIONS:
Behavioral: Brief Behavioral Therapy for Insomnia (BBTI) — Participants will receive evidence-based 'Brief Behavioral Therapy for Insomnia' (BBTI), tailored to meet the needs of former football players. BBTi is a brief, efficacious treatment that focuses on modifying behaviors, rather than cognitive domains. The treatment emphasizes education, motivational tools, and specific behavioral recommendations (e.g., restricting time in bed) and will be administered through weekly phone calls with a trained sleep interventionist over 4-weeks.

SUMMARY:
This pilot study is focused on estimating the impact of a tele-sleep intervention on patient-centered outcomes relevant to former football players, including a) sleep duration, quality, and daytime impairment; b) pain, pain catastrophizing, physical and emotional functioning; c) mood; d) quality of life, with the longer-term goal to evaluate the impact on cardiovascular health risk. The evidence-based 'Brief Behavioral Therapy for Insomnia' (BBTI) will be utilized and tailored it to meet the needs of former football players.

This pilot work will serve as the foundation for a larger, future clinical trial that utilizes a durable approach for improving sleep health with potential influence pain and quality of life as well as future studies to evaluate the implementation and scalability of BBTI in novel populations.

DETAILED DESCRIPTION:
The investigators will plan to enroll 40 participants. Players will be recruited from the Harvard Football Players Health Study cohort from across the US via email and telephone invitations. Following screening, if the participant is eligible and interested, they may consent to enroll in the study. Participants will receive evidence-based 'Brief Behavioral Therapy for Insomnia' (BBTI), tailored to meet the needs of former football players. BBTi is a brief, efficacious treatment that focuses on modifying behaviors, rather than cognitive domains. The treatment emphasizes education, motivational tools, and specific behavioral recommendations (e.g., restricting time in bed). BBTI has been previously delivered remotely and this intervention will be delivered by phone by sleep interventionists including trained social workers, psychologists, and nurse practitioners. Participants will complete an intake session with their interventionist followed by a 'treatment session' a week later wherein the interventionist will provide education about sleep regulation and create an individualized schedule of sleep/wake times for the participant. This will be followed by 3 brief weekly check-in calls to review progress, address questions and concerns, and adjust the behavioral treatment plan as the participant progresses. The participant will complete a daily sleep diary throughout the intervention to inform the treatment. Participants will also complete baseline, endpoint and follow-up questionnaires to assess outcomes and intervention acceptability and feasibility. Participants will receive compensation for their participation.

ELIGIBILITY:
Inclusion criteria

* Able to communicate clearly in English
* Have a digital device with reliable internet access
* Sub-clinical insomnia (Insomnia Severity Index, score >7, sub-clinical threshold insomnia)
* Able to give informed consent

Exclusion criteria

* Prior participation in behavioral therapy for insomnia
* Self-reported circadian phase irregularity/delay, including regular shift work
* Previously diagnosed Narcolepsy, bipolar disorder or other major psychiatric disorders
* Active alcohol abuse (Alcohol Use Disorders Identification Test, AUDIT-C ≥4) or drug abuse (Drug Abuse Screening Test, DAST-2 ≥1)
* Current severe major depressive disorder (Patient Health Questionnaire-8, PHQ-8, score ≥20)
* Use of seizure medication or seizure within the past 10 years
* Untreated, previously diagnosed moderate to severe sleep apnea or excessive daytime sleepiness (defined by Epworth sleepiness scale score ≥16) with a self-reported sleep duration (>6 hours)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-09-07 (Actual)

PRIMARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance, 8b Endpoint | Week 4
  PROMIS Sleep Disturbance measures self-reported sleep quality and associated daytime functioning during the past seven days. The measure includes 8-items with higher scores indicating greater sleep disturbance. The minimum score is 8 and the maximum score is 40. Item responses are combined to yield a T-score with a population mean of 50 and standard deviation of 10.

SECONDARY OUTCOMES:
PROMIS Sleep Disturbance, 8b Follow-up | Week 12
  PROMIS Sleep Disturbance measures self-reported sleep quality and associated daytime functioning during the past seven days. The measure includes 8-items with higher scores indicating greater sleep disturbance. The minimum score is 8 and the maximum score is 40. Item responses are combined to yield a T-score with a population mean of 50 and standard deviation of 10.
PROMIS Sleep Impairment, 8a Endpoint | Week 4
  PROMIS Sleep Impairment measures self-reported perceptions of alertness, sleepiness, and tiredness during usual waking hours, and the perceived functional impairments during wakefulness associated with sleep problems or impaired alertness during the past seven days. The measure includes 8-items with higher scores indicating greater sleep impairment. The minimum score is 8 and the maximum score 40. Item responses are combined to yield a T-score with a population mean of 50 and standard deviation of 10.
PROMIS Sleep Impairment, 8a Follow-up | Week 12
  PROMIS Sleep Impairment measures self-reported perceptions of alertness, sleepiness, and tiredness during usual waking hours, and the perceived functional impairments during wakefulness associated with sleep problems or impaired alertness during the past seven days. The measure includes 8-items with higher scores indicating greater sleep disturbance. The minimum score is 8 and the maximum score 40. Item responses are combined to yield a T-score with a population mean of 50 and standard deviation of 10.
Response to treatment (baseline to endpoint) | Week 0 vs. Week 4
  Previous 'Brief Behavioral Treatment for Insomnia' interventions have defined response to treatment as a change in the PSQI score of ≥3 points (Buysse, 2011). The PSQI, or the Pittsburgh Sleep Quality Index, is a validated instrument which assesses self-reported sleep quality and disturbances over a 1-month interval. The minimum score is 0 and maximum score is 21. Higher scores indicate worse sleep quality.
Response to treatment (baseline to follow-up) | Week 0 vs. Week 12
  Previous 'Brief Behavioral Treatment for Insomnia' interventions have defined response to treatment as a change in the PSQI score of ≥3 points (Buysse, 2011). The PSQI, or the Pittsburgh Sleep Quality Index, is a validated instrument which assesses self-reported sleep quality and disturbances over a 1-month interval. The minimum score is 0 and maximum score is 21. Higher scores indicate worse sleep quality.
Remission of poor sleep symptoms (baseline to endpoint) | Week 0 vs. Week 4
  Previous 'Brief Behavioral Treatment for Insomnia' interventions have defined remission as the response criterion (change in the PSQI score of ≥3 points) plus a final PSQI score <5 (Buysse, 2011). The PSQI, or the Pittsburgh Sleep Quality Index, is a validated instrument which assesses self-reported sleep quality and disturbances over a 1-month interval. The minimum score is 0 and maximum score is 21. Higher scores indicate worse sleep quality.
Remission of poor sleep symptoms (baseline to follow-up) | Week 0 vs. Week 12
  Previous 'Brief Behavioral Treatment for Insomnia' interventions have defined remission as the response criterion (change in the PSQI score of ≥3 points) plus a final PSQI score <5 (Buysse, 2011). The PSQI, or the Pittsburgh Sleep Quality Index, is a validated instrument which assesses self-reported sleep quality and disturbances over a 1-month interval. The minimum score is 0 and maximum score is 21. Higher scores indicate worse sleep quality.
PROMIS Pain intensity, 3a (Endpoint) | Week 4
  PROMIS Pain intensity 3a is a self-report measure that assesses how much a person hurts (intensity or severity) in the past 7 days. The measure includes three items rating pain from "Had no pain" = 1 to "Very severe" = 5, therefore the response range is 3-15 with higher scores indicating greater pain intensity. Item responses are combined to yield a T-score with population mean of 50 and standard deviation of 10.
PROMIS Pain intensity, 3a (Follow-up) | Week 12
  PROMIS Pain intensity 3a is a self-report measure that assesses how much a person hurts (intensity or severity) in the past 7 days. The measure includes three items rating pain from "Had no pain" = 1 to "Very severe" = 5, therefore the response range is 3-15 with higher scores indicating greater pain intensity. Item responses are combined to yield a T-score with population mean of 50 and standard deviation of 10.
PROMIS Pain interference, 8a (Endpoint) | Week 4
  PROMIS Pain interference 8a assesses self-reported consequences of pain on relevant aspects of one's life in the past 7 days.
  The measure includes 8-items rating pain from "Not at all" = 1 to "Very much" = 5, therefore the response range is 8-40 with higher scores indicating greater pain interference. Item responses are combined to yield a standardized T-score with a mean of 50, and a standard deviation of 10.
PROMIS Pain interference, 8a (Follow-up) | Week 12
  PROMIS Pain interference 8a assesses self-reported consequences of pain on relevant aspects of one's life in the past 7 days.
  The measure includes 8-items rating pain from "Not at all" = 1 to "Very much" = 5, therefore the response range is 8-40 with higher scores indicating greater pain interference. Item responses are combined to yield a standardized T-score with a mean of 50, and a standard deviation of 10.
Insomnia Severity Index, ISI (Endpoint) | Week 4
  The Insomnia Severity Index is a 7-item self-report questionnaire assessing the nature, severity, and impact of insomnia in the last month. A 5-point Likert scale is used to rate each item (e.g., 0 = no problem; 4 = very severe problem), yielding a total score ranging from 0 to 28. The total score is interpreted as follows: absence of insomnia (0-7); sub-threshold insomnia (8-14); moderate insomnia (15-21); and severe insomnia (22-28).
Insomnia Severity Index, ISI (Follow-up) | Week 12
  The Insomnia Severity Index is a 7-item self-report questionnaire assessing the nature, severity, and impact of insomnia in the last month. A 5-point Likert scale is used to rate each item (e.g., 0 = no problem; 4 = very severe problem), yielding a total score ranging from 0 to 28. The total score is interpreted as follows: absence of insomnia (0-7); sub-threshold insomnia (8-14); moderate insomnia (15-21); and severe insomnia (22-28).

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Bertisch, MD, MPH, Principal Investigator — Assistant Professor in Medicine, Physician/Clinical Investigator
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No